CLINICAL TRIAL: NCT02574104
Title: Generalizing TESTPILOT-NICU: Transportable Enhanced Simulation Technologies for Pre-Implementation Limited Operations Testing in Neonatal Intensive Care Units
Brief Title: Generalizing TESTPILOT to New Single Family Room NICUs
Acronym: TESTPILOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jesse Bender, Neonatologist, Women and Infants Hospital of Rhode Island
Other Study IDs: 792397-1
Record Dates: First submitted 2015-10-07; First posted 2015-10-12 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Patient Safety; Organizational Change
Keywords: Intensive Care Units, Neonatal; Patient simulation; Interdisciplinary Communication; Human factors; Hazard Analysis and Critical Control Points

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (15):
- Institution 1: McGill University Health Center NICU staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Complete
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 2: Rochester University Medical Center NICU staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Complete
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 3: Parkland Memorial Hospital NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Complete
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 4: Eastern Maine Medical Center NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Active
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 5: Brigham and Women's Hospital NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Active
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 6: Centre hospitalier universitaire Sainte-Justine NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Active
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 7: Golisano Children's Hospital of Southwest Florida NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Preparing
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 8: Florida Hospital for Children NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Preparing
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 9: Memorial Hospital of South Bend NICU Staff
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  STATUS: Pending
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 10: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 11: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 12: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 13: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 14: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients
- Institution 15: recruiting
  Simulate a functional NICU prior to moving patients to preserve safety at transition
  Interventions: Other: Simulate a functional NICU prior to moving patients

INTERVENTIONS:
Other: Simulate a functional NICU prior to moving patients — Test translation of care paradigms in the new environment a priori. Invest significant time and resources into scenario design, staffing, preparing and orchestration the simulations. 80-160 staff participate in simulations, discover and resolve latent safety threats

SUMMARY:
Complex service interventions are neither smooth nor easy in any transitioning healthcare facility. Simulations performed in the new environment reinforce patient safety by uncovering safety threats, enabling their correction, and orienting hospital staff. This study expands upon patient safety successes at several institutions to measurably enhance patient safety at upcoming new inpatient facilities.

DETAILED DESCRIPTION:
Prior to opening the nation's largest single family room NICU in 2009, Women & Infants Hospital developed TESTPILOT: Transportable Enhanced Simulation Technologies for Pre-Implementation Limited Operations Testing. The investigators simulated a functional NICU. 164 latent safety threats (LST) were identified without exposing a single neonate to risk. Practical changes were made to a) verbal and written communication protocols, b) admissions workflows, c) rapid team responses, d) family centered care e) scripting, f) facilities, g) supplies and equipment, and h) staffing and training issues.

"Generalizing TESTPILOT" studies how learnable and applicable this simulation-based methodology is at other institutions. Six institutions have successfully implemented TESTPILOT-NICU as of 2015. The investigators hypothesize implementations will succeed across a spectrum of care delivery structures, simulation experience and magnitudes of culture change, resulting in a broad blueprint for integrating simulation into transitioning healthcare services. Our goals include:

1. Share lessons learned and support local simulation teams in their preparations;
2. Quantitatively demonstrate improvement in system readiness and staff preparedness at each institution
3. Assess saturation of latent safety threats over successive TESTPILOT implementations, resulting in a blueprint for similar transitions.

During Phase I the investigators standardized, refined and validated survey instruments with NICU staff and process experts. Phase II includes implementation of TESTPILOT at 15 institutions over three years. The Principal Investigator recruits each institution and guides them through the methodology, typically lasting six to eight months. Each institution's Co-Investigator and core simulation team recruits local staff for simulation, LST discovery and resolution, and survey completion.

ELIGIBILITY:
Inclusion Criteria:

* NICUs transitioning during the study period will be recruited.
* Active NICU staff at each institution will be encouraged to participate without regard to age, gender, race, pregnancy or health status.
* The participants will be a representative sample of the overall staff, which includes primarily women in most NICUs.

Exclusion Criteria:

* Institutions unable to commit resources for simulation preparation, latent safety threat correction, or study reporting requirements

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Institutions building a new single family room or hybrid Neonatal Intensive Care Unit (NICU)
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-10 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Cumulative Latent Safety Threats (LST) discovered | Two months leading up to transition
  LSTs are discovered during simulations, documented during debriefings, fed back to workflow committees for corrective action, and solutions may be retested in subsequent simulations

SECONDARY OUTCOMES:
Average change in system readiness | Baseline (12-8 weeks prior to move), post-TESTPILOT (6-4 weeks prior), post-workshop (10 days prior) and post-transition (4-8 weeks post)
  Clinical staff will document the readiness improvement trajectory of 24 key NICU processes with 6-point Likert responses to surveys in these time frames
Average change in staff preparedness | Baseline (12-8 weeks prior to move), post-TESTPILOT (6-4 weeks prior), post-workshop (10 days prior) and post-transition (4-8 weeks post)
  Clinical staff will document the improvement trajectory of their preparedness to perform these same 24 key NICU processes with 6-point Likert responses to surveys in the time frames
Qualitative review of successes and challenges | 90 minute focus group discussion three months after transition
  Structured team discussion on successes and ongoing challenges

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Bender, MD, Principal Investigator — Women & Infants Hospital
Locations (1):
- Women & Infants Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Summary level data will be made available to other researchers

REFERENCES:
- [Background] Bender J, Shields R, Kennally K. Transportable enhanced simulation technologies for pre-implementation limited operations testing: neonatal intensive care unit. Simul Healthc. 2011 Aug;6(4):204-12. doi: 10.1097/SIH.0b013e3182183c0b. PMID 21546863
- [Background] Kobayashi L, Shapiro MJ, Sucov A, Woolard R, Boss RM 3rd, Dunbar J, Sciamacco R, Karpik K, Jay G. Portable advanced medical simulation for new emergency department testing and orientation. Acad Emerg Med. 2006 Jun;13(6):691-5. doi: 10.1197/j.aem.2006.01.023. Epub 2006 Apr 24. PMID 16636356
- [Background] Kaji AH, Bair A, Okuda Y, Kobayashi L, Khare R, Vozenilek J. Defining systems expertise: effective simulation at the organizational level--implications for patient safety, disaster surge capacity, and facilitating the systems interface. Acad Emerg Med. 2008 Nov;15(11):1098-103. doi: 10.1111/j.1553-2712.2008.00209.x. Epub 2008 Aug 20. PMID 18717649
- [Background] Villamaria FJ, Pliego JF, Wehbe-Janek H, Coker N, Rajab MH, Sibbitt S, Ogden PE, Musick K, Browning JL, Hays-Grudo J. Using simulation to orient code blue teams to a new hospital facility. Simul Healthc. 2008 Winter;3(4):209-16. doi: 10.1097/SIH.0b013e31818187f3. PMID 19088665
- [Background] Bender GJ. In situ simulation for systems testing in newly constructed perinatal facilities. Semin Perinatol. 2011 Apr;35(2):80-3. doi: 10.1053/j.semperi.2011.01.007. PMID 21440815